CLINICAL TRIAL: NCT00122824
Title: Duloxetine Hydrochloride 60 mg or 120 mg Once Daily Compared With Placebo in Patients With Generalized Anxiety Disorder.
Brief Title: Duloxetine Compared With Placebo in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5075; F1J-MC-HMBR
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine hydrochloride
Drug: placebo

SUMMARY:
This is a clinical trial assessing duloxetine compared with placebo in patients who have generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients at least 18 years of age

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating duloxetine or have previously been treated with duloxetine
* Patient diagnosed with major depressive disorder within the past 6 months
* Patient diagnosed with panic disorder, post-traumatic stress disorder, or an eating disorder within the past year
* History of alcohol or any psychoactive substance abuse or dependence within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2004-06; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To assess duloxetine 120 mg once daily is superior to placebo in the treatment of GAD, defined as statistically greater reduction on the mean change anxiety symptoms as measured by the HAMA total score.

SECONDARY OUTCOMES:
Self-reported anxiety symptomatology;Pain;Quality of Life;Clinical Global Improvement;HAMA factor scores

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-285-4559 or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Cincinnati, Ohio, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Oulu, Finland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Bourg-en-Bresse, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Berlin, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Paarl, South Africa
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Barcelona, Spain
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Uppsala, Sweden

REFERENCES:
- [Derived] Sheehan DV, Harnett-Sheehan K, Spann ME, Thompson HF, Prakash A. Assessing remission in major depressive disorder and generalized anxiety disorder clinical trials with the discan metric of the Sheehan disability scale. Int Clin Psychopharmacol. 2011 Mar;26(2):75-83. doi: 10.1097/YIC.0b013e328341bb5f. PMID 21102344
- [Derived] Sheehan DV, Meyers AL, Prakash A, Robinson MJ, Swindle RW, Russell JM, Mallinckrodt CH. The relationship between functional outcomes and the treatment of anxious and painful somatic symptoms in patients with generalized anxiety disorder. Curr Med Res Opin. 2008 Sep;24(9):2457-66. doi: 10.1185/03007990802293643. Epub 2008 Jul 24. PMID 18662492
- [Derived] Hartford JT, Endicott J, Kornstein SG, Allgulander C, Wohlreich MM, Russell JM, Perahia DG, Erickson JS. Implications of pain in generalized anxiety disorder: efficacy of duloxetine. Prim Care Companion J Clin Psychiatry. 2008;10(3):197-204. doi: 10.4088/pcc.v10n0304. PMID 18615176
- [Derived] Koponen H, Allgulander C, Erickson J, Dunayevich E, Pritchett Y, Detke MJ, Ball SG, Russell JM. Efficacy of duloxetine for the treatment of generalized anxiety disorder: implications for primary care physicians. Prim Care Companion J Clin Psychiatry. 2007;9(2):100-7. doi: 10.4088/pcc.v09n0203. PMID 17607331
- [Derived] Allgulander C, Hartford J, Russell J, Ball S, Erickson J, Raskin J, Rynn M. Pharmacotherapy of generalized anxiety disorder: results of duloxetine treatment from a pooled analysis of three clinical trials. Curr Med Res Opin. 2007 Jun;23(6):1245-52. doi: 10.1185/030079907X182202. Epub 2007 Apr 25. PMID 17559726
- [Derived] Endicott J, Russell JM, Raskin J, Detke MJ, Erickson J, Ball SG, Marciniak M, Swindle RW. Duloxetine treatment for role functioning improvement in generalized anxiety disorder: three independent studies. J Clin Psychiatry. 2007 Apr;68(4):518-24. doi: 10.4088/jcp.v68n0405. PMID 17474806
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com